CLINICAL TRIAL: NCT04384978
Title: Development of Serious Games and Physical Activities Instructed by a Social Robot for Improving the Well-being of Elderly Individuals With Alzheimer's Disease and Dementia
Brief Title: Socially Assistive Robots for Interaction With Older Adults With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DreamFace Technologies, LLC (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Mohammad Mahoor, Founder and CEO, DreamFace Technologies, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-001; R44AG066439-01 (NIH)
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A 12-month pilot study will be comprised of two groups of people diagnosed with mild Alzheimer's disease and related dementia for a total of 80 senior subjects. Subjects will be randomly assigned to two groups: Group 1 users will play games with and administered by Ryan, 2-3 times a week and 30-minutes per day. Group 2 (Active Control Group) will play solitary games and activities but will have to interaction with Ryan. The team will measure the changes and improvement in the social/emotional well-being of these two groups and eventual changes in the cognitive/memory functions of elderly people living in the similar environment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Control Group: Group 2 users will play solitary games (word puzzles) and activities but will have no interaction with Ryan.
  Interventions: Behavioral: Play Solitary Games Without a Social Robot
- Active Group (Experimental): Active Group: Group 1 users will play games with and administered by Ryan, 2-3 times a week and 30-minutes per day.
  Interventions: Behavioral: Play Serious Games with a Social Robot (Ryan)

INTERVENTIONS:
Behavioral: Play Serious Games with a Social Robot (Ryan) — Active Group: Game play and physical activities with Ryan, a socially assistive robot developed at DreamFace Technologies,LLC.
  Arms: Active Group
Behavioral: Play Solitary Games Without a Social Robot — Control Group: Group 2 will play solitary games (e.g., word puzzles) and activities but will have no interaction with Ryan.
  Arms: Control Group

SUMMARY:
A 12-month pilot study will be comprised of two groups of people diagnosed with mild Alzheimer's disease and related dementia for a total of 80 senior subjects. Subjects will be randomly assigned to two groups: Group 1 users will play games with and administered by Ryan, 2-3 times a week and 30-minutes per day. Group 2 (Active Control Group) will play solitary games and activities but will have to interaction with Ryan. The team will measure the changes and improvement in the social/emotional well-being of these two groups and eventual changes in the cognitive/memory functions of elderly people living in the similar environment.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 65 years
* Early Alzheimer's disease and related dementia diagnosed by a qualified provider
* Saint Louis University Mental Status (SLUMS) score between 10 and 25
* Resident of assisted living facility for at least one month prior and for the duration of the study
* Deemed conditioned enough to participate in physical activities after a wellness check
* Verbal skill to interact
* Participant or Legal decision

Exclusion Criteria:

Aggressive behavior

* Diagnosed with severe dementia or memory loss
* Acute physical illness that impairs ability to participate
* Patients with serious comorbidity, tumors and other diseases casually related to cognitive impairment
* History of alcohol or drug abuse, head trauma, psychoactive substance use and other causes of memory impairment
* Significant sensory impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2022-03-06 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eaton Senior Communities, Lakewood, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Active Group
Started | 4 | 18
Completed | 0 | 18
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Active Group | Total
Number analyzed (Participants) | 4 | 18 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 4 | 18 | 22
Age, Continuous [Mean (Standard Deviation); unit: Year] | 80.20 (5.44) | 76.2 (6.11) | 77.7 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 1 | 6 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 4 | 15 | 19
  Race/Ethnicity: Hispanic | 0 | 2 | 2
  Race/Ethnicity: Asian | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 18 | 22
The Saint Louis University Mental Status (SLUMS) [Mean (Standard Deviation); unit: units on a scale] — The SLUMS exam tests several cognitive domains, as listed below: Verbal memory (13 points) Attention/concentration (5 points) Visuospatial/constructional abilities (5 points). The scale range is between 0-30 and the higher the score the better.
  For individuals who have completed a high school education, the SLUMS score structure is as follows: 27-30: Indicates regular cognitive function. 21-26: Indicates mild cognitive impairment. 1-20: Indicates dementia.
  units on a scale | 19.12 (4.10) | 21.12 (3.20) | 20.45 (3.34)

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive/Memory Ability
Description: Participants will complete the Saint Louis University Mental Status (SLUMS) test, a screening method for Alzheimer's and other dementia. Scores range from 0 to 30. Scores of 27 to 30 are considered normal in a person with a high school education. Scores between 21 and 26 suggest a mild neurocognitive disorder. Scores between 0 and 20 indicate dementia.
Time Frame: assessed at baseline (week 1), week 4, and 8. Week 8 reported.
Population: The participants did not complete the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Group | Control Group
Number analyzed (Participants) | 18 | 0
score on a scale | 23.75 (3.45) |

ADVERSE EVENTS:
Time Frame: The adverse events were monitored and assessed at the participant level (up to 10 weeks) throughout the study. As a result, no adverse events were reported during the study period.
Description: No adverse event was reported.
Arm/Group | Control Group | Active Group
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/18
Other Adverse Events (participants affected / at risk) | 0/4 | 0/18

LIMITATIONS AND CAVEATS:
The study was conducted right after COVID-19 restrictions were lifted. The main limitation was that some potential subjects had medical constraints or concerns and did not want to participate. Additionally, poor internet connections in some senior care facilities limited the ability to converse with the robot.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT04384978/Prot_SAP_000.pdf